CLINICAL TRIAL: NCT01653236
Title: Pilot Study to Determine the Efficacy and Safety of Combining Boceprevir With Peginterferon Alfa-2b and Ribavirin in the Treatment-naive Patients Infected With Genotype 4 Chronic Hepatitis C Infection
Brief Title: Boceprevir With Peginterferon Alfa-2b and Ribavirin in the Treatment-naive Patients Infected With Genotype 4 Chronic Hepatitis C Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mostafa Ibrahim, Vice President, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3034-108
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Genotype 4 Chronic Hepatitis C Infection
MeSH Terms: interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm B (Experimental): 48 weeks of peginterferon alfa-2b and ribavirin Plus Boceprevir 800 mg
  Interventions: Drug: Boceprevir; Drug: Peginterferon alfa-2b; Drug: ribavirin
- Control Arm (Active Comparator): 48 weeks of peginterferon alfa-2b and ribavirin
  Interventions: Drug: Peginterferon alfa-2b; Drug: ribavirin

INTERVENTIONS:
Drug: Boceprevir
  Arms: Experimental Arm B
Drug: Peginterferon alfa-2b
Drug: ribavirin

SUMMARY:
Hypothesis Combination of Boceprevir with Ribavirin in treatment-naïve patients with genotype 4 chronic hepatitis C infection will increase the proportion of patients achieving sustained viral response compared to standard treatment alone.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to assess the efficacy and safety of Boceprevir 800 mg three times per day (TID) orally (PO) (hereafter called Boceprevir) in combination with peginterferon alfa-2b 1.5 μg/kg once per week (QW) subcutaneously (SC) plus weight-based dosing (WBD) of ribavirin (800 to 1400 mg/day) compared to standard of care (SOC) (therapy with peginterferon alfa-2b (PEG)+ribavirin (RBV) WBD) in previously untreated adult subjects with chronic hepatitis C (CHC) genotype 4 infection.

Primary Trial Objectives:

- The primary efficacy objective of this study is to assess the efficacy of Boceprevir in combination with PEG 1.5 μg/kg QW SC plus WBD of RBV (800 to 1400 mg/day) compared to the efficacy of SOC (therapy with PEG+RBV WBD) in the Control Arm in previously untreated adult subjects with CHC genotype 4 infection

ELIGIBILITY:
* Ages Eligible for Study: 18 Years and older
* Genders Eligible for Study: Both

Inclusion Criteria:

* Subject must be more than 18 years of age.
* Subject's weight must be more than 40 kg and less than 125 kg.
* Subject and subject's partner must each agree to use acceptable methods of contraception for at least 2 weeks prior to Day 1 and continue until at least 6 months after last dose of study medication, or longer if dictated by local regulations.
* Subjects must be willing to give written informed consent for the trial and for the pharmacogenetic testing.
* Subjects who are unwilling to provide written informed consent for pharmacogenetic testing may be included in the trial; however, pharmacogenetic samples must not be obtained.
* Subject must have previously documented CHC genotype 4 infection.
* Subjects with other or mixed genotypes are not eligible. The HCV-RNA result obtained from the central laboratory at the screening visit must confirm genotype 4 infection and be more10,000 IU per mL Previously untreated patients with Pegylated interferon
* Subject must have a liver biopsy or fibrotest and fibroscan with histology consistent with CHC and no other etiology.

Exclusion Criteria:

* Subject who is coinfected with the human immunodeficiency virus (HIV) or hepatitis B virus.
* Prior treatment with interferon, ribavirin and/or investigational agent for hepatitis C.
* Prior treatments with herbal remedies with known hepatotoxicity are exclusionary.
* All herbal remedies used for hepatitis C treatment must be discontinued before Day 1.
* Treatment with any investigational drug within 30 days of the screening visit in this trial.
* Subject who received any of the following medication(s) within 2 weeks prior to the Day 1 visit that are highly dependent on CYP3A4.5 for clearance, and for which elevated plasma concentrations are associated with serious and or life-threatening events such as: orally administered midazolam, pimozide, amiodarone, flecainide, propafenone, quinidine and ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine).
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 72 Weeks
  The primary efficacy objective of this study is to assess the efficacy of Boceprevir in combination with PEG 1.5 μg/kg QW SC plus WBD of RBV (800 to 1400 mg/day) compared to the efficacy of SOC (therapy with PEG+RBV WBD) in the Control Arm in previously untreated adult subjects with CHC genotype 4 infection

SECONDARY OUTCOMES:
Week 8 Response | 8 weeks
  1. Assess the number of patients who achieved SVR after achieving undetectable or ≥2 log reduction of HCV RNA level at treatment week 8;
12 Weeks response | 12 weeks
  Assess the number of patients who achieved SVR after achieving undetectable or ≥2 log reduction of HCV RNA level at treatment week 12
IL-28B polymorphism | 72 Weeks
  To evaluate the effect of IL-28B polymorphism (CC,CT,TT) alleles on the viral kinetic response after the addition of Boceprevir

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

REFERENCES:
- [Background] Poordad F, McCone J Jr, Bacon BR, Bruno S, Manns MP, Sulkowski MS, Jacobson IM, Reddy KR, Goodman ZD, Boparai N, DiNubile MJ, Sniukiene V, Brass CA, Albrecht JK, Bronowicki JP; SPRINT-2 Investigators. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1195-206. doi: 10.1056/NEJMoa1010494. PMID 21449783